CLINICAL TRIAL: NCT01533506
Title: Compassionate Use of Stiripentol in Intractable Epilepsy Due to Dravet Syndrome
Brief Title: Stiripentol in Dravet Syndrome
Status: No longer available | Type: Expanded Access
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Elaine C. Wirrell, Consultant, Mayo Clinic
Other Study IDs: 12-000690
Record Dates: First submitted 2012-02-09; First posted 2012-02-15 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Dravet Syndrome
Keywords: treatment with stiripentol
MeSH Terms: conditions — Epilepsies, Myoclonic | interventions — stiripentol

INTERVENTIONS:
Drug: stiripentol — Stiripentol up to 30 mg/kg/day to control seizures
  Other Names: Diacomit

SUMMARY:
The patient has failed all other available agents and has intractable epilepsy due to Dravet Syndrome. Stiripentol is highly efficacious in Dravet Syndrome. The overall goals of therapy with Stiripentol are primarily to significantly reduce the frequency and severity of seizures.

ELIGIBILITY:
Inclusion Criteria:

* Genetic diagnosis of Dravet syndrome with intractable seizures despite failing all available medications for seizures

Min Age: 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2012-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Wirrell, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States